CLINICAL TRIAL: NCT01486238
Title: Pegaptanib for Retinal Edema Secondary to Diabetic Vascular Disease(Preserve) Study
Acronym: PRESERVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valley Retina Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRESERVE
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema
MeSH Terms: interventions — pegaptanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVMac q6 Arm (Experimental): Patients assigned to IVMac q6 will receive a total of 4 intravitreal Macugen® injections administered at 6week intervals beginning on Day 0 and ending at Week 18. Macugen® injection will be administered as described in the package insert.
  Interventions: Drug: Macugen® pegaptanib sodium
- IVMac q4 Arm (Experimental): Patients assigned to IVMac q4 will receive a total of 6 intravitreal Macugen® injections administered at 4 week intervals beginning on Day 0 and ending at Week 20. Macugen® injection will be administered as described in the package insert.
  Interventions: Drug: Macugen® pegaptanib sodium

INTERVENTIONS:
Drug: Macugen® pegaptanib sodium — Patients assigned to either arm (IVMac q4 and IVMac q6) will receive 0.3 milligrams (mg) of pegaptanib sodium delivered by intravitreal injection administered.
  Patients assigned to IVMac q4 will receive a total of 6 intravitreal Macugen® injections administered at 4 week intervals beginning on Day 0 and ending at Week 20. Patients assigned to IVMac q6 will receive a total of 4 intravitreal Macugen® injections administered at 6 week intervals beginning on Day 0 and ending at Week 18. Each Macugen® injection will be administered as described in the package insert.
  Other Names: Macugen® (pegaptanib sodium)

SUMMARY:
Intravitreal injections of pegaptanib every 4 weeks will be efficacious in treating Diabetic Macular Edema (DME), as compared to injections every 6 weeks.

DETAILED DESCRIPTION:
This is a 24 week clinical study which will be double-masked. Subjects will be randomly assigned 2:1 to Macugen® every 4 weeks (IVMac q4 arm) or Macugen® every 6 weeks (IVMac q6 arm). If both eyes are eligible, then one eye will be randomized into the trial. Fellow eyes of patients with two eligible eyes will be monitored and treated with standard clinical care. If sufficient fellow eyes are treated, this will provide an internal control group for direct comparison of the Macugen® treated study eyes versus the fellow eyes. Both study eyes and fellow eyes will be assessed in the same fashion at every time point during this study.

Each site is to have at least one Unmasked investigator to perform the study injections and one Masked investigator to perform study evaluations and assess adverse events. Roles cannot be reversed after study treatment for a given subject has begun.

Patients assigned to IVMac q4 will receive a total of 6 intravitreal Macugen® injections administered at 4 week intervals beginning on Day 0 and ending at Week 20. Patients assigned to IVMac q6 will receive a total of 4 intravitreal Macugen® injections administered at 6 week intervals beginning on Day 0 and ending at Week 18. Each Macugen® injection will be administered as described in the package insert.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have macular edema that involves the center of the macula with corresponding leakage on fluorescein angiogram.
2. Foveal thickness of at least 250 microns (OCT center point thickness), with a standard deviation of the center point of <10%, an OCT signal strength of > 5, and properly drawn ILM and RPE borders.
3. Best corrected distance visual acuity in the study eye must 137 be a letter score between 70 and 20 inclusive (20/40 to 20/400 Snellen equivalents).
4. Clear ocular media and adequate pupillary dilatation to permit good quality stereoscopic fundus photography.
5. Intraocular pressure (IOP) of 21 mmHg or less (local anti-hypertensive medication of any duration permitted).
6. The treating ophthalmologist should be comfortable that focal laser (direct and grid as needed) can be deferred for at least 18 weeks in the study eye, even though focal laser is indicated.
7. Type I, or Type II diabetic subjects, of both genders, and aged 18 years.
8. Women must be using effective contraception, be post-menopausal for at least 12 months prior to trial entry, or surgically sterile. All women of childbearing potential must have a negative serum pregnancy test at baseline and negative urine pregnancy tests immediately prior to each injection and use two effective forms of contraception during the trial and for at least 60 days following the last dose of pegaptanib sodium.
9. Ability to provide written informed consent.
10. Ability to return for all study visits.

Exclusion Criteria:

1. Eyes in which panretinal photocoagulation is needed now or is likely to be needed within the next 6 months.
2. Eyes that have active PDR with high risk characteristics (HRC) as defined by the DRS:

   1. Mild neovascularization of the disc (NVD) of at least 1/3 disc area as shown in standard photograph 10A of the DRS.
   2. Moderate neovascularization of the retina elsewhere (NVE) of at least 1/2 disc area as shown in standard photograph 7 of the DRS.
3. Presence of any abnormality that is likely to confound assessment of visual acuity improvement in eyes in which macular edema resolves, or improves, such as non-perfusion for >1 disc area involving the foveal avascular zone, epiretinal membrane associated with signs of contraction and/or significant opacification, or presence of chorioretinal atrophy involving the center of the macula.
4. Vitreomacular traction determined clinically and/or by OCT, which, in the investigator's opinion, contributes to the macular edema (or causes associated foveal detachment), and would preclude improvement with pegaptanib sodium
5. Any other cause of macular edema such as vitreous extension, or entrapment to anterior segment wound, or any retinal vein occlusion involving the macula.
6. Any subfoveal hard exudates, or RPE atrophy; or any present evidence, or past documentation of a foveal cyst (by fundus examination, FA or OCT).
7. Previous treatment with intravitreal corticosteroids in the study eye within 3 months of Day 0 visit.
8. Previous treatment with intravitreal anti-angiogenic drugs in the study eye within 3 months of Day 0 visit.
9. Previous PRP laser treatment in the study eye within 90 days of Day 0 visit.
10. Subjects who have received YAG laser or peripheral retinal cryoablation or laser retinopexy (for retinal tears only), or focal photocoagulation within the previous 16 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Gonzalez, Dr., Principal Investigator — Valley Retina Institute
Locations (1):
- Valley Retina Institute,PA, McAllen, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited from a single medical clinic (Valley Retina Institute), and randomly assigned 2:1 to Macugen® every 4 weeks (IVMac q4 arm) or Macugen® every 6 weeks (IVMac q6 arm). If both eyes are eligible, then one eye will be randomized into the trial.
Pre-assignment Details: All enrolled patients must have DME in one or both eyes. In patients with both eyes that meet criteria, only 1 eye will be considered eligible. All fellow eyes in these patients will be treated according to standard clinical guidelines.
Period: Overall Study
Arm/Group | IVMac q6 Arm | IVMac q4 Arm
Started | 23 | 49
Completed | 21 | 43
Not Completed | 2 | 6
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: In the IVMac q6 Arm, 23 subjects started the study. Two (2) subjects withdrew early. For this reason data from the 21 remaining subjects was used.
  In the IVMac q4 Arm, 49 subjects started the study. 6 subjects were lost in this arm - 2 died, 1 withdrew, & 3 were lost to follow-up. For this reason data from the 43 remaining subjects was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | IVMac q6 Arm | IVMac q4 Arm | Total
Number analyzed (Participants) | 21 | 43 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 41 | 55
  >=65 years | 7 | 2 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 62 (30) | 62.5 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 21 | 30
  Male | 12 | 22 | 34
Region of Enrollment [Number; unit: participants]
  United States | 21 | 43 | 64

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Gain Two or More Lines in Best Corrected Visual Acuity(BCVA) Score in the Study Eye Compared With Baseline.
Description: The primary efficacy outcome measure is the proportion of subjects who gain two or more lines in BCVA score in the Study Eye compared with baseline at 24 weeks. The BCVA is to be measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol.
Time Frame: 24 weeks
Population: Proportion of subjects who gain two or more lines BCVA was calculated.
Measure: Number; unit: participants
Arm/Group | IVMac q6 Arm | IVMac q4 Arm
Number analyzed (Participants) | 21 | 43
participants | 3 | 18

2. Secondary Outcome: Mean Change From Baseline at Week 24 in Central Foveal Thickness
Description: Optical Coherence Tomography (OCT) will be used to assess the central foveal thickness of each patient. The mean change from baseline to week 24 will be calculated for each patient.
Time Frame: 24 Weeks
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Subjects Requiring Macular Laser Treatment at Week 12 and Week 24.
Description: There is a possibility that some subjects may not respond to the study treatment to which they have been assigned. Macular laser treatment is considered an alternative treatment for retinal edema. A lower proportion of subjects requiring macular laser treatment would indicate a superior treatment regimen.
  This will be assessed at week 12, and again at week 24.
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | IVMac q6 Arm | IVMac q4 Arm
Serious Adverse Events (participants affected / at risk) | 3/23 | 12/49
Other Adverse Events (participants affected / at risk) | 0/21 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVMac q6 Arm (N=23) | IVMac q4 Arm (N=49)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Non study drug related
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) — Not related to study drug
Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1) — not related to study drug
Pneumonia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — not related to study drug
Left Foot Abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — not related to study drug
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — not related to study drug
Neovascularization of the Iris (Eye disorders) | 0 (0) | 1 (1)
Severe Retrosternal Chest Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — not related to study drug
Septicemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — not related to study drug
Uncontrolled High Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1) — not related to study drug
Ischemic Neuropathy left eye (Eye disorders) | 1 (1) | 1 (1) — not related to study drug
Unknown Death (Investigations) | 0 (0) | 1 (1) — cause of death was unknown upon completion of the trial
Unknown Death (Investigations) | 0 (0) | 1 (1) — cause of death was unknown at the completion of the trial
Left Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — not related to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No